CLINICAL TRIAL: NCT03689829
Title: A Parallel-design Phase 1 Study to Assess Safety, Tolerability and Pharmacokinetics/Exposure Following Different Single Dose Levels of MOR106 (Administered Subcutaneously or Intravenously) in Healthy Male Subjects (Randomized, Open-label), and in Subjects With Moderate to Severe Atopic Dermatitis (Randomized, Placebo-controlled, Double-blind, Repeated Subcutaneous Dosing Over 12 Weeks)
Brief Title: A Study to Test Safety, Tolerability, and the Way the Body Absorbs, Distributes, and Gets Rid of a Study Drug Called MOR106, in Healthy Subjects and in Patients With Moderate to Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: MOR106 clinical development in atopic dermatitis was stopped for futility
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MOR106-CL-102; 2018-000357-44 (EudraCT Number)
Record Dates: First submitted 2018-09-20; First posted 2018-09-28 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Healthy; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Masking Description: Part 1 - randomized open label. Part 2 and Part 3 - randomized double blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- MOR106 Single Dose A, i.v. infusion, Part 1 (Experimental): A single dose of MOR106 will be administered by i.v. infusion.
  Interventions: Drug: MOR106
- MOR106 Single Dose B, s.c. injection, Part 1 (Experimental): A single dose of MOR106 will be administered by s.c. injection.
  Interventions: Drug: MOR106
- MOR106 Single Dose C, s.c. injection, Part 1 (Experimental): A single dose of MOR106 will be administered by s.c. injection.
  Interventions: Drug: MOR106
- MOR106 Single Dose D, s.c. injection, Part 1 (Experimental): A single dose of MOR106 will be administered by s.c. injection.
  Interventions: Drug: MOR106
- MOR106 Repeated Doses E, s.c. injection, Part 2 (Experimental): Repeated doses of MOR106 will be administered by s.c. injection with a loading dose on the first day of administration.
  Interventions: Drug: MOR106
- Placebo s.c.injection, Part 2 (Placebo Comparator): Corresponding Placebo will be administered by s.c. injection.
  Interventions: Drug: Placebo
- MOR106 Repeated Doses F, s.c. injection, Part 3 (Experimental): Repeated doses of MOR106 will be administered by s.c. injection with a loading dose on the first day of administration.
  Interventions: Drug: MOR106
- Placebo s.c.injection, Part 3 (Placebo Comparator): Corresponding Placebo will be administered by s.c. injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MOR106 — The active pharmaceutical drug substance of MOR106 is a human immunoglobulin gamma-1 (IgG1) monoclonal antibody that binds with a high apparent affinity to human interleukin-17C (IL-17C).
  Arms: MOR106 Repeated Doses E, s.c. injection, Part 2; MOR106 Repeated Doses F, s.c. injection, Part 3; MOR106 Single Dose A, i.v. infusion, Part 1; MOR106 Single Dose B, s.c. injection, Part 1; MOR106 Single Dose C, s.c. injection, Part 1; MOR106 Single Dose D, s.c. injection, Part 1
Drug: Placebo — Corresponding placebo s.c. injections.
  Arms: Placebo s.c.injection, Part 2; Placebo s.c.injection, Part 3

SUMMARY:
The clinical study consists of three parts:

* Part 1 with healthy volunteers.
* Part 2 and Part 3 including subjects with moderate to severe atopic dermatitis (a skin disease).

For Part 1 the main goal of the study is to compare the safety, tolerability, and exposure of administration of the test drug via an injection in a skin layer just under the surface (subcutaneous), to administration of the test drug into the vein (intravenous).

For Part 2 and Part 3 the main goal of the study is to assess the safety and tolerability of administration of the test drug via an injection in a skin layer just under the surface (subcutaneous) during 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Male between 18-50 years of age (extremes included), on the day of signing the informed consent form (ICF).
* Subjects between 65-88 kg (extremes included) with a body mass index (BMI) between 18-30 kg/m², inclusive.
* Judged to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and screening laboratory profile prior to the initial investigation medicinal product (IMP) administration.

Part 2 and Part 3:

* Male or female between 18-65 years of age (extremes included), on the day of signing ICF.
* A BMI between 18-30 kg/m², inclusive.
* Diagnosis of AD for at least one year since first diagnosis as per Hanifin and Rajka Criteria.
* EASI ≥ 12 at screening and ≥ 16 at the baseline visit (Day 1 predose)
* ≥ 10% BSA of AD involvement at screening.
* IGA score ≥ 3 (on 0-4 IGA scale).
* Willingness to use an additive free, basic, bland emollient twice daily for at least seven days before the baseline visit and throughout the study.
* Subject is a candidate for systemic therapy and is not responding adequately or has a contraindication to topical corticosteroids (TCS) and / or topical calcineurin inhibitors (TCI), per investigator's judgment.

Exclusion Criteria:

Part 1, Part 2 and Part 3:

* Known hypersensitivity to IMP ingredients as determined by the investigator (such as, but not limited to, anaphylaxis requiring hospitalization).
* Prior treatment with MOR106.
* Any concurrent illness, condition, disability, or clinically significant abnormality (including laboratory tests, ≥ New York Heart Association Classification (NYHA) III/IV) or clinically significant illness in the three months prior to initial IMP administration that, in the investigator's opinion, represents a safety risk for the subject's participation in the study, may affect the interpretation of clinical safety or efficacy data, or may prevent the subject from safely completing the assessments required by the protocol.
* History of, or current immunosuppressive condition.

In addition for Part 2 and 3:

* Active chronic or acute skin infection requiring treatment with systemic (oral, sc or iv) antibiotics, antivirals or antifungals within 4 weeks of baseline, or clinical signs of infective eczema within 1 week before baseline (Day 1 pre-dose).
* Having used any of the following treatments:

  i) Exposure to a biologic therapy for AD. ii) Immunosuppressive/ immunomodulating drugs (e.g. systemic corticosteroids, cyclosporine, mycophenolate-mofetil, interferon-γ (IFN-γ), azathioprine, methotrexate, etc.) within 4 weeks of baseline. iii) Phototherapy (ultraviolet (UVB) or Psoralen Ultraviolet A [PUVA]) for AD within four weeks of baseline. iv) Treatment with TCS or TCI within two weeks before the baseline visit. v) Treatment with biologics (for non-AD indications) within five half-lives (if known) or 12 weeks prior to baseline visit, whichever is longer. vi) Regular use (more than two visits per week) of a tanning booth/parlor within four weeks of the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
The number of incidents of Treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), serious adverse events (SAEs) and discontinuations due to Adverse Events (AEs) Part 1. | From study drug administration until Day 50 postdose or early discontinuation (ED) visit
  To evaluate the safety and tolerability of single doses of MOR106 administered s.c. in comparison to i.v.
The number of incidents of Treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), serious adverse events (SAEs) and discontinuations due to Adverse Events (AEs) Part 2. | From study drug administration until Day 197 postdose or early discontinuation (ED) visit
  To evaluate the safety and tolerability of multiple doses of MOR106 administered s.c.
The number of incidents of Treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), serious adverse events (SAEs) and discontinuations due to Adverse Events (AEs) Part 3. | From study drug administration until Day 155 postdose or early discontinuation (ED) visit
  To evaluate the safety and tolerability of multiple doses of MOR106 administered s.c.
AUC ratio between s.c. and i.v. dosing (area under the plasma concentration-time curve) Part 1. | Between Day 1 study period and Day 50 postdose or early discontinuation (ED) visit
  To determine the relative bioavailability following sc route of administration.
Area under the serum concentration-time curve from time zero to infinity (AUC0-inf) Part 1. | Between Day 1 study period and Day 50 postdose or early discontinuation (ED) visit
  To characterize the pharmacokinetics (PK) of MOR106.
Terminal elimination half-life (t1/2) Part 1. | Between Day 1 study period and Day 50 postdose or early discontinuation (ED) visit
  To characterize the PK of MOR106.
Maximum observed plasma concentration (Cmax) Part 1. | Between Day 1 study period and Day 50 postdose or early discontinuation (ED) visit
  To characterize the PK of MOR106.

SECONDARY OUTCOMES:
Occurrence of anti-drug antibodies (ADA) Part 1. | From baseline through Day 50 postdose or early discontinuation (ED) visit
  To monitor the occurrence of ADA after single administrations of MOR106.
Occurrence of anti-drug antibodies (ADA) Part 2. | From baseline through Day 197 postdose or early discontinuation (ED) visit
  To monitor the occurrence of ADA after multiple administrations of MOR106.
Occurrence of anti-drug antibodies (ADA) Part 3. | From baseline through Day 155 postdose or early discontinuation (ED) visit
  To monitor the occurrence of ADA after multiple administrations of MOR106.
MOR106 serum concentrations after multiple s.c. administrations Part 2. | Between Day 1 study period and Day 197 postdose or early discontinuation (ED) visit
  Steady-state will be assessed using MOR106 serum concentrations.
MOR106 serum concentrations after multiple s.c. administrations Part 3. | Between Day 1 study period and Day 155 postdose or early discontinuation (ED) visit
  Steady-state will be assessed using MOR106 serum concentrations.
Percent change in Eczema Area and Severity Index (EASI) Part 2. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of EASI score. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Percent change in Eczema Area and Severity Index (EASI) Part 3. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of EASI score. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve ≥50% overall improvement in Eczema Area and Severity Index (EASI) score Part 2. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of EASI score. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve ≥50% overall improvement in Eczema Area and Severity Index (EASI) score Part 3. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of EASI score. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Time to first response of Eczema Area and Severity Index (EASI) improvement with 50% Part 2. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of EASI score. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Time to first response of Eczema Area and Severity Index (EASI) improvement with 50% Part 3. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of EASI score. The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve ≥75% and ≥90% improvement in Eczema Area and Severity Index (EASI) Part 2. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of EASI score,The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve ≥75% and ≥90% improvement in Eczema Area and Severity Index (EASI) Part 3. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of EASI score,The EASI score ranges are between 0 (no eczema) and 72. Higher values represent a worse outcome.
Proportion of subjects who achieve an Investigators' Global Assessment (IGA) score of 0 or 1 Part 2. | at Day 85 visit
  To assess the efficacy of MOR106 by use of IGA score, an assessment scale to determine severity of AD and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe) score. Higher values represent a worse outcome.
Proportion of subjects who achieve an Investigators' Global Assessment (IGA) score of 0 or 1 Part 3. | at Day 85 visit
  To assess the efficacy of MOR106 by use of IGA score, an assessment scale to determine severity of AD and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe) score. Higher values represent a worse outcome.
Proportion of subjects who achieve an Investigators' Global Assessment (IGA) score reduction of ≥2 Part 2. | at Day 85 visit
  To assess the efficacy of MOR106 by use of IGA score, an assessment scale to determine severity of AD and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe) score. Higher values represent a worse outcome.
Proportion of subjects who achieve an Investigators' Global Assessment (IGA) score reduction of ≥2 Part 3. | at Day 85 visit
  To assess the efficacy of MOR106 by use of IGA score, an assessment scale to determine severity of AD and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe) score. Higher values represent a worse outcome.
Percent change in Scoring Atopic Dermatitis (SCORAD) score Part 2. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of SCORAD.The SCORAD evaluates the extent of atopic dermatitis and ranges between 0 and 103. Higher values represent a worse outcome.
Percent change in Scoring Atopic Dermatitis (SCORAD) score Part 3. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of SCORAD.The SCORAD evaluates the extent of atopic dermatitis and ranges between 0 and 103. Higher values represent a worse outcome.
Absolute and percent change in body surface area (BSA), Patient Oriented Eczema Measure (POEM) score Part 2. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of POEM. The POEM is calculated by summing the score of each question resulting in a maximum score of 28 and a minimum score of 0.
Absolute and percent change in body surface area (BSA), Patient Oriented Eczema Measure (POEM) score Part 3. | From baseline to Day 85
  To assess the efficacy of MOR106 by use of POEM. The POEM is calculated by summing the score of each question resulting in a maximum score of 28 and a minimum score of 0.
Weekly change from baseline in Pruritus Numeric Rating Scale (NRS) Part 2. | From screening until Day 197 or early discontinuation (ED) visit twice daily
  To assess the efficacy of MOR106 by NRS. An 11-point (0 - 10) scale will be used to assess itch (pruritus). 0 being 'no itch' and 10 being the 'worst itch imaginable'.
Weekly change from baseline in Pruritus Numeric Rating Scale (NRS) Part 3. | From screening until Day 155 or early discontinuation (ED) visit twice daily
  To assess the efficacy of MOR106 by NRS. An 11-point (0 - 10) scale will be used to assess itch (pruritus). 0 being 'no itch' and 10 being the 'worst itch imaginable'.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Timmis, MB CHB, Study Director — Galapagos NV
Locations (15):
- Germany (6):
  - Klinikum Augsburg Süd, Augsburg
  - Municipal Hospital Dessau, Dessau
  - University Hospital Carl Gustav Carus, Dresden
  - University Hospital Erlangen, Department of Dermatology, Erlangen
  - Medical Faculty University Clinic Magdeburg, University dermatology clinic, Magdeburg
  - Vest Clinic, Department of Dermatology and Allergy, Recklinghausen
- Spain (4):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia
- Arensia, Kapitanivka, Ukraine
- United Kingdom (4):
  - MEU, Manchester
  - MeDiNova North London, Northwood
  - MeDiNova East London, Romford
  - MeDiNova South London, Sidcup